CLINICAL TRIAL: NCT01889784
Title: Evaluation of Acute Effect of Phototherapy With Light Emitting Diode (LED) on Muscle and Pulmonary Oxygen Consumption in Patients With Diabetes Mellitus
Brief Title: Acute Effect of Phototherapy With Light Emitting Diode (LED) on Muscle and Pulmonary Oxygen Consumption on Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aparecida Maria Catai (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor-Investigator, Aparecida Maria Catai, PhD, Universidade Federal de Sao Carlos
Organization: Universidade Federal de Sao Carlos (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 13573013.1.0000.5504
Record Dates: First submitted 2013-06-05; First posted 2013-06-28 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes mellitus, type 2; phototherapy; physical exercise; oxygen consumption; arterial blood pressure; heart rate; baroreflex sensitivity; cardiovascular autonomic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Individuals with diabetes mellitus (phototherapy 150J) (Other): The intervention of this study is phototherapy through light emitting diode (LED) and dose of 150J each muscle. The Effective-LED or Placebo-LED will be applied in femoral quadriceps and triceps surae muscles bilaterally before constant-load exercise tests in bike. Each individual will perform two tests with Effective-LED and two tests with Placebo-LED randomly allocated. Evaluations will be completed in 4 days in total, respecting 14 days of rest to ensure the long washout phototherapy.
  Interventions: Device: Phototherapy through light emitting diode (LED) - 150J; Device: Placebo phototherapy - 150J
- Health individuals - 150J (phototherapy 150J) (Other): The intervention of this study is phototherapy through light emitting diode (LED) and dose of 150J each muscle. The Effective-LED or Placebo-LED will be applied in femoral quadriceps and triceps surae muscle bilaterally before constant-load exercise tests in bike. Each individual will perform two tests with Effective-LED and two tests with Placebo-LED randomly allocated. Evaluations will be completed in 4 days in total, respecting 14 days of rest to ensure the long washout phototherapy.
  Interventions: Device: Phototherapy through light emitting diode (LED) - 150J; Device: Placebo phototherapy - 150J
- Individuals with diabetes mellitus (phototherapy 300J) (Other): The intervention of this study is phototherapy through light emitting diode (LED) with 300J. The Effective-LED or Placebo-LED will be applied in femoral quadriceps and triceps surale muscles bilaterally before constant-load exercise tests in bike. Each individual will perform two tests with Effective-LED and two tests with Placebo-LED randomly allocated. Evaluations will be completed in 4 days in total, respecting 14 days of rest to ensure the long washout phototherapy.
  Interventions: Device: Phototherapy through light emitting diode (LED) - 300J; Device: Placebo phototherapy - 300J
- Health individuals (phototherapy 300J) (Other): The intervention of this study is phototherapy through light emitting diode (LED). The Effective-LED or Placebo-LED will be applied in femoral quadriceps and triceps surae muscle bilaterally before constant-load exercise tests in bike. Each individual will perform two tests with Effective-LED and two tests with Placebo-LED randomly allocated. Evaluations will be completed in 4 days in total, respecting 14 days of rest to ensure the long washout phototherapy.
  Interventions: Device: Phototherapy through light emitting diode (LED) - 300J; Device: Placebo phototherapy - 300J

INTERVENTIONS:
Device: Phototherapy through light emitting diode (LED) - 150J — The near-infrared radiation by light emitting diode (LED) will be performed with a cluster multi-diode arranged in an array of 34x18 cm containing 50 LEDs (GaAlAs, 850 nm). The phototherapy will be applied bilaterally on femoral quadriceps and triceps surae muscles during 40 seconds with 3J of total energy for each diode and 150 J of total energy delivery to muscle. Neither subject nor evaluators will known if LED was effective or placebo during data collection. A hidden button in the LED device is employed to ensure the double-blind procedure. This button allows selecting placebo or effective emission of near-infrared radiation while the time display is working. This button will be selected by a researcher who just participated of randomization procedure and LED application and had no access to data collection.
  Arms: Health individuals - 150J (phototherapy 150J); Individuals with diabetes mellitus (phototherapy 150J)
Device: Placebo phototherapy - 150J — The near-infrared radiation by light emitting diode (LED) will be performed with a cluster multi-diode arranged in an array of 34x18 cm containing 50 LEDs (GaAlAs, 850 nm). The phototherapy will be applied bilaterally on femoral quadriceps and triceps surae muscles during 40 seconds with 3J of total energy for each diode and 150 J of total energy delivery to muscle. Neither subject nor evaluators will known if LED was effective or placebo during data collection. A hidden button in the LED device is employed to ensure the double-blind procedure. This button allows selecting placebo or effective emission of near-infrared radiation while the time display is working. This button will be selected by a researcher who just participated of randomization procedure and LED application and had no access to data collection.
  Arms: Health individuals - 150J (phototherapy 150J); Individuals with diabetes mellitus (phototherapy 150J)
Device: Phototherapy through light emitting diode (LED) - 300J — The near-infrared radiation by light emitting diode (LED) will be performed with a cluster multi-diode arranged in an array of 34x18 cm containing 50 LEDs (GaAlAs, 850 nm). The phototherapy will be applied bilaterally on femoral quadriceps and triceps surae muscles during 80 seconds with 6J of total energy for each diode and 300 J of total energy delivery to muscle. Neither subject nor evaluators will known if LED was effective or placebo during data collection. A hidden button in the LED device is employed to ensure the double-blind procedure. This button allows selecting placebo or effective emission of near-infrared radiation while the time display is working. This button will be selected by a researcher who just participated of randomization procedure and LED application and had no access to data collection.
  Arms: Health individuals (phototherapy 300J); Individuals with diabetes mellitus (phototherapy 300J)
Device: Placebo phototherapy - 300J — The near-infrared radiation by light emitting diode (LED) will be performed with a cluster multi-diode arranged in an array of 34x18 cm containing 50 LEDs (GaAlAs, 850 nm). The phototherapy will be applied bilaterally on femoral quadriceps and triceps surae muscles during 80 seconds with 6J of total energy for each diode and 300 J of total energy delivery to muscle. Neither subject nor evaluators will known if LED was effective or placebo during data collection. A hidden button in the LED device is employed to ensure the double-blind procedure. This button allows selecting placebo or effective emission of near-infrared radiation while the time display is working. This button will be selected by a researcher who just participated of randomization procedure and LED application and had no access to data collection.
  Arms: Health individuals (phototherapy 300J); Individuals with diabetes mellitus (phototherapy 300J)

SUMMARY:
The purpose of this study is to determine the phototherapy may be adjuvant to exercise to improve muscular efficiency and increase aerobic capacity. We hypothesized that phototherapy adjuvant with physical exercise may be benefit to populations with Diabetes mellitus that have impairment in cardiopulmonary fitness and low oxygen uptake peak values (VO2peak) in exercise tests. Two doses will be tested 150J and 300J.

Additionally, this study aims to evaluate the effect of phototherapy previously applied to the exercise on the cardiovascular coupling. We hypothesize that phototherapy previously applied to the exercise will result in the increase baroreflex sensitivity (increased coherence and gain and decreased phase), promoting the improvement of the cardiovascular autonomic control and cardiovascular coupling in diabetic subjects. Two doses will be tested 150J and 300J.

ELIGIBILITY:
Inclusion Criteria:

* overt coronary disease
* sedentary
* Clinical diagnosis of diabetes mellitus
* Free of diabetes mellitus to participate of control group

Exclusion Criteria:

* autonomic neuropathy
* Smoking
* anemia
* alcoholism
* disability conditions precluding exercise

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change in muscle oxygen uptake after phototherapy and placebo phototherapy with light emitting diode (LED) - 150J | Change in muscle oxygen uptake after phototherapy and placebo phototherapy initial, 2 weeks, 4 weeks and 6 weeks
  20 men with diabetes mellitus will receive effective-phototherapy (cluster multi-diode containing 50 LEDs applied for 40 seconds over muscle quadriceps bilaterally) or Placebo-phototherapy using the same device and procedures. Effective and placebo phototherapy will be performed 2 times each and the sequence will be random, with 14 days of rest between evaluations. The therapies will be applied 10 minutes before dynamic physical exercise of constant workload and moderate intensity to evaluate the phototherapy effect in muscle oxygen uptake evaluated through near-infrared spectroscopy (NIRS) (Oxymon system, Artinis Medical Systems, Netherlands). The optode of NIRS will be fixed on quadriceps muscle in the right side.
Change in muscle oxygen uptake after phototherapy and placebo phototherapy with light emitting diode (LED) - 300J | Change in muscle oxygen uptake after phototherapy and placebo phototherapy initial, 2 weeks, 4 weeks and 6 weeks
  20 men with diabetes mellitus will receive effective-phototherapy (cluster multi-diode containing 50 LEDs applied for 80 seconds over muscle quadriceps bilaterally) or Placebo-phototherapy using the same device and procedures. Effective and placebo phototherapy will be performed 2 times each and the sequence will be random, with 14 days of rest between evaluations. The therapies will be applied 10 minutes before dynamic physical exercise of constant workload and moderate intensity to evaluate the phototherapy effect in muscle oxygen uptake evaluated through near-infrared spectroscopy (NIRS) (Oxymon system, Artinis Medical Systems, Netherlands). The optode of NIRS will be fixed on quadriceps muscle in the right side.

SECONDARY OUTCOMES:
Change in pulmonary oxygen uptake after phototherapy and placebo phototherapy with light emitting diode (LED) - 150J | Change in pulmonary oxygen uptake after phototherapy and placebo phototherapy initial, 2 weeks, 4 weeks and 6 weeks
  20 men with diabetes mellitus and 20 health men will receive effective-phototherapy (cluster multi-diode containing 50 LEDs applied for 40 seconds over muscle quadriceps bilaterally) or Placebo-phototherapy using the same device and procedures. Effective and placebo phototherapy will be performed 2 times each and the sequence will be random, with 14 days of rest between evaluations. The therapies will be applied 10 minutes before dynamic physical exercise of constant workload and moderate intensity to evaluate the phototherapy effect in pulmonary oxygen uptake evaluated through metabolic unit (CPX/D, MedGraphics, St. Paul, Minnesota, USA) continuously collected breath-by-breath.
Change in pulmonary oxygen uptake after phototherapy and placebo phototherapy with light emitting diode (LED) - 300J | Change in pulmonary oxygen uptake after phototherapy and placebo phototherapy initial, 2 weeks, 4 weeks and 6 weeks
  20 men with diabetes mellitus and 20 health men will receive effective-phototherapy (cluster multi-diode containing 50 LEDs applied for 80 seconds over muscle quadriceps bilaterally) or Placebo-phototherapy using the same device and procedures. Effective and placebo phototherapy will be performed 2 times each and the sequence will be random, with 14 days of rest between evaluations. The therapies will be applied 10 minutes before dynamic physical exercise of constant workload and moderate intensity to evaluate the phototherapy effect in pulmonary oxygen uptake evaluated through metabolic unit (CPX/D, MedGraphics, St. Paul, Minnesota, USA) continuously collected breath-by-breath.
Change in baroreflex sensitivity after phototherapy and placebo phototherapy with light emitting diode (LED) - 150J | Time Frame: Change in pulmonary oxygen uptake after phototherapy and placebo phototherapy initial, 2 weeks, 4 weeks and 6 weeks
  20 men with diabetes mellitus and 20 health men will receive effective-phototherapy (cluster multi-diode containing 50 LEDs applied for 40 seconds over muscle quadriceps bilaterally) or Placebo-phototherapy using the same device and procedures. Effective and placebo phototherapy will be performed 2 times each and the sequence will be random, with 14 days of rest between evaluations. The therapies will be applied 10 minutes before dynamic physical exercise of constant workload and moderate intensity to evaluate the phototherapy effect in baroreflex sensitivity evaluated through pulse plethysmograph (Finometer PRO, Finapres Medical Systems, The Netherlands).
Change in baroreflex sensitivity after phototherapy and placebo phototherapy with light emitting diode (LED) - 300J | Time Frame: Change in pulmonary oxygen uptake after phototherapy and placebo phototherapy initial, 2 weeks, 4 weeks and 6 weeks
  20 men with diabetes mellitus and 20 health men will receive effective-phototherapy (cluster multi-diode containing 50 LEDs applied for 80 seconds over muscle quadriceps bilaterally) or Placebo-phototherapy using the same device and procedures. Effective and placebo phototherapy will be performed 2 times each and the sequence will be random, with 14 days of rest between evaluations. The therapies will be applied 10 minutes before dynamic physical exercise of constant workload and moderate intensity to evaluate the phototherapy effect in baroreflex sensitivity evaluated through pulse plethysmograph (Finometer PRO, Finapres Medical Systems, The Netherlands).

OTHER OUTCOMES:
Change in arterial blood pressure after phototherapy and placebo phototherapy with light emitting diode (LED) - 150J | Change in arterial blood pressure after phototherapy and placebo phototherapy initial, 2 weeks, 4 weeks and 6 weeks
  20 men with diabetes mellitus will receive effective-phototherapy (cluster multi-diode containing 50 LEDs applied for 40 seconds over muscle quadriceps bilaterally) or Placebo-phototherapy using the same device and procedures. Effective and placebo phototherapy will be performed 2 times each and the sequence will be random, with 14 days of rest between evaluations. The therapies will be applied 10 minutes before dynamic physical exercise of constant workload and moderate intensity to evaluate the phototherapy effect in arterial blood pressure evaluated continuously through pulse plethysmograph (Finometer PRO, Finapres Medical Systems, The Netherlands)
Change in arterial blood pressure after phototherapy and placebo phototherapy with light emitting diode (LED) - 300J | Change in arterial blood pressure after phototherapy and placebo phototherapy initial, 2 weeks, 4 weeks and 6 weeks
  20 men with diabetes mellitus will receive effective-phototherapy (cluster multi-diode containing 50 LEDs applied for 80 seconds over muscle quadriceps bilaterally) or Placebo-phototherapy using the same device and procedures. Effective and placebo phototherapy will be performed 2 times each and the sequence will be random, with 14 days of rest between evaluations. The therapies will be applied 10 minutes before dynamic physical exercise of constant workload and moderate intensity to evaluate the phototherapy effect in arterial blood pressure evaluated continuously through pulse plethysmograph (Finometer PRO, Finapres Medical Systems, The Netherlands)
Change in glucose and lactate concentrations after phototherapy and placebo phototherapy with light emitting diode (LED) - 150J | Change in glucose and lactate concentrations after phototherapy and placebo phototherapy initial, 2 weeks, 4 weeks and 6 weeks
  20 men with diabetes mellitus will receive effective-phototherapy (cluster multi-diode containing 50 LEDs applied for 40 seconds over muscle quadriceps bilaterally) or Placebo-phototherapy using the same device and procedures. Effective and placebo phototherapy will be performed 2 times each and the sequence will be random, with 14 days of rest between evaluations. The therapies will be applied 10 minutes before dynamic physical exercise of constant workload and moderate intensity to evaluate the phototherapy effect in glucose and lactate concentrations. Blood samples will be collected by puncturing ear lobe before and 10 minutes after each exercise test had been concluded and will be processed with glucose and lactate analyser (YSI 2300 STAT PLUS - Yellow Springs Instruments - Yellow Springs, USA)
Change in glucose and lactate concentrations after phototherapy and placebo phototherapy with light emitting diode (LED) - 300J | Change in glucose and lactate concentrations after phototherapy and placebo phototherapy initial, 2 weeks, 4 weeks and 6 weeks
  20 men with diabetes mellitus will receive effective-phototherapy (cluster multi-diode containing 50 LEDs applied for 80 seconds over muscle quadriceps bilaterally) or Placebo-phototherapy using the same device and procedures. Effective and placebo phototherapy will be performed 2 times each and the sequence will be random, with 14 days of rest between evaluations. The therapies will be applied 10 minutes before dynamic physical exercise of constant workload and moderate intensity to evaluate the phototherapy effect in glucose and lactate concentrations. Blood samples will be collected by puncturing ear lobe before and 10 minutes after each exercise test had been concluded and will be processed with glucose and lactate analyser (YSI 2300 STAT PLUS - Yellow Springs Instruments - Yellow Springs, USA)
Change in heart rate after phototherapy and placebo phototherapy with light emitting diode (LED) - 150J | Change in heart rate after phototherapy and placebo phototherapy initial, 2 weeks, 4 weeks and 6 weeks
  20 men with diabetes mellitus will receive effective-phototherapy (cluster multi-diode containing 50 LEDs applied for 40 seconds over muscle quadriceps bilaterally) or Placebo-phototherapy using the same device and procedures. Effective and placebo phototherapy will be performed 2 times each and the sequence will be random, with 14 days of rest between evaluations. The therapies will be applied 10 minutes before dynamic physical exercise of constant workload and moderate intensity to evaluate the phototherapy effect in heart rate evaluated continuously through pulse plethysmograph (Finometer PRO, Finapres Medical Systems, The Netherlands)
Change in heart rate after phototherapy and placebo phototherapy with light emitting diode (LED) - 300J | Change in heart rate after phototherapy and placebo phototherapy initial, 2 weeks, 4 weeks and 6 weeks
  20 men with diabetes mellitus will receive effective-phototherapy (cluster multi-diode containing 50 LEDs applied for 80 seconds over muscle quadriceps bilaterally) or Placebo-phototherapy using the same device and procedures. Effective and placebo phototherapy will be performed 2 times each and the sequence will be random, with 14 days of rest between evaluations. The therapies will be applied 10 minutes before dynamic physical exercise of constant workload and moderate intensity to evaluate the phototherapy effect in heart rate evaluated continuously through pulse plethysmograph (Finometer PRO, Finapres Medical Systems, The Netherlands)

CONTACTS AND LOCATIONS:
Overall Officials: Aparecida M Catai, pHD, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Universidade Federal de São Carlos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The individual data is shared with each patient. The data will be published in journal with impact in the area, but the personal information of the participants will not be uncovered.

REFERENCES:
- [Background] Vieira WH, Ferraresi C, Perez SE, Baldissera V, Parizotto NA. Effects of low-level laser therapy (808 nm) on isokinetic muscle performance of young women submitted to endurance training: a randomized controlled clinical trial. Lasers Med Sci. 2012 Mar;27(2):497-504. doi: 10.1007/s10103-011-0984-0. Epub 2011 Aug 26. PMID 21870127
- [Background] Leal Junior EC, Lopes-Martins RA, Vanin AA, Baroni BM, Grosselli D, De Marchi T, Iversen VV, Bjordal JM. Effect of 830 nm low-level laser therapy in exercise-induced skeletal muscle fatigue in humans. Lasers Med Sci. 2009 May;24(3):425-31. doi: 10.1007/s10103-008-0592-9. Epub 2008 Jul 23. PMID 18649044
- [Background] Paolillo FR, Milan JC, Aniceto IV, Barreto SG, Rebelatto JR, Borghi-Silva A, Parizotto NA, Kurachi C, Bagnato VS. Effects of infrared-LED illumination applied during high-intensity treadmill training in postmenopausal women. Photomed Laser Surg. 2011 Sep;29(9):639-45. doi: 10.1089/pho.2010.2961. Epub 2011 Jul 12. PMID 21749263
- [Background] Leal Junior EC, Lopes-Martins RA, Rossi RP, De Marchi T, Baroni BM, de Godoi V, Marcos RL, Ramos L, Bjordal JM. Effect of cluster multi-diode light emitting diode therapy (LEDT) on exercise-induced skeletal muscle fatigue and skeletal muscle recovery in humans. Lasers Surg Med. 2009 Oct;41(8):572-7. doi: 10.1002/lsm.20810. PMID 19731300
- [Background] Ihsan FR. Low-level laser therapy accelerates collateral circulation and enhances microcirculation. Photomed Laser Surg. 2005 Jun;23(3):289-94. doi: 10.1089/pho.2005.23.289. PMID 15954817
- [Background] Vladimirov YA, Osipov AN, Klebanov GI. Photobiological principles of therapeutic applications of laser radiation. Biochemistry (Mosc). 2004 Jan;69(1):81-90. doi: 10.1023/b:biry.0000016356.93968.7e. PMID 14972023
- [Background] Bauer TA, Reusch JE, Levi M, Regensteiner JG. Skeletal muscle deoxygenation after the onset of moderate exercise suggests slowed microvascular blood flow kinetics in type 2 diabetes. Diabetes Care. 2007 Nov;30(11):2880-5. doi: 10.2337/dc07-0843. Epub 2007 Aug 3. PMID 17675540
- [Background] Wilkerson DP, Poole DC, Jones AM, Fulford J, Mawson DM, Ball CI, Shore AC. Older type 2 diabetic males do not exhibit abnormal pulmonary oxygen uptake and muscle oxygen utilization dynamics during submaximal cycling exercise. Am J Physiol Regul Integr Comp Physiol. 2011 Mar;300(3):R685-92. doi: 10.1152/ajpregu.00479.2010. Epub 2010 Dec 22. PMID 21178129
- [Derived] Francisco Cde O, Beltrame T, Ferraresi C, Parizotto NA, Bagnato VS, Borghi Silva A, Benze BG, Porta A, Catai AM. Evaluation of acute effect of light-emitting diode (LED) phototherapy on muscle deoxygenation and pulmonary oxygen uptake kinetics in patients with diabetes mellitus: study protocol for a randomized controlled trial. Trials. 2015 Dec 15;16:572. doi: 10.1186/s13063-015-1093-3. PMID 26666374